CLINICAL TRIAL: NCT01301144
Title: Sensitivity and Specificity of Oral Urea Breath Testing for Presumptive Diagnosis and Treatment Response in Pulmonary Tuberculosis in Bamako, Mali
Brief Title: Oral Urea Breath Testing for Diagnosis and Treatment Response in Pulmonary Tuberculosis
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911106; 11-I-N106
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-03-30

CONDITIONS: Tuberculosis; Urea Breath Test
Keywords: Tuberculosis; Urea Breath Test
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Tuberculosis is a disease of the lungs caused by the bacteria Mycobacterium tuberculosis (M. tuberculosis). The most popular and least expensive tool used to detect the presence of the tuberculosis bacteria is called sputum smears, which is a lab test used to look for bacteria in the sputum via a microscope. However, the test s results are not always accurate, and the test cannot determine if the bacteria will be resistant to standard tuberculosis treatments. The most sensitive test currently available is called sputum culture, in which a sputum sample is used to check for the growth of tuberculosis bacteria. However, this test takes at least a month to produce accurate results, and requires expensive equipment that is not available in many countries where M. tuberculosis is found.
* The urea breath test (UBT) has been used to detect infection with Helicobacter pylori, a bacteria associated with stomach ulcers, by testing individual breath samples. Researchers are interested in determining whether breath samples can also be used to detect the presence of M. tuberculosis in the lungs of subjects with tuberculosis, and to see if tuberculosis treatments are successful.

Objectives:

- To assess the sensitivity and specificity of urea breath testing in the diagnosis and treatment response of pulmonary tuberculosis.

Eligibility:

* Individuals at least 18 years of age who either have been diagnosed with tuberculosis or are healthy volunteers with no past history of tuberculosis.
* The study will be conducted in Bamako, Mali.

Design:

* This study will involve three groups: two pilot groups of individuals who have already been diagnosed with tuberculosis, and a primary study group of both healthy volunteers and individuals who have been diagnosed with tuberculosis.
* Participants will be screened with a physical examination and medical history, as well as blood, sputum, stool, and urine samples.
* First pilot group (one visit):
* Participants should not eat, drink, or smoke for at least 1 hour prior to the UBT test.
* Participants will provide a baseline exhaled air sample, and then will receive the UBT test, which involves a dose of Pranactin -Citric dissolved in water. Additional exhaled air samples will be collected at eight time points (10, 20, 45, 60, 90, 120, 180, and 240 minutes after the dose).
* Second pilot group (one or two visits):
* Participants should not eat, drink, or smoke for at least 1 hour prior to the UBT test.
* Participants will provide a baseline exhaled air sample, and then will receive the UBT test. Half of the participants will receive a dose of bismuth (Pepto-Bismol) prior to collection of air samples to see how this affects the results of the UBT test. Additional exhaled air samples will be collected at three time points specified by the study researchers.
* On the following day, participants will return for a second visit to provide three more exhaled air samples.
* Primary study group (five visits for participants with tuberculosis, two visits for healthy volunteers):
* All participants will have two visits, following the procedures given for the second pilot group. Half will receive a dose of bismuth prior to collection of air samples.
* Participants with tuberculosis will have three additional visits (days 6, 10, and 16 following the first study visit) to provide additional sputum and exhaled air samples to monitor the progress of tuberculosis treatment.

DETAILED DESCRIPTION:
Tuberculosis (TB) is a disease that affects the population worldwide, with 9 million people being infected every year. It is associated with high rates of mortality and morbidity. Reports show that a person dies from tuberculosis every 20 seconds worldwide. Current diagnostic techniques are either inadequate at detecting TB cases with precision, or they are time consuming, expensive, and require laboratory equipment not available in developing countries, where the disease is endemic. Furthermore, rates of multi-drug-resistant (MDR) TB are estimated to be over 5 percent of the incident cases globally and extremely drug-resistant (XDR) TB rates are on the rise. These statistics highlight the need for new and improved diagnostic tools for TB, as well as biomarkers that can quickly detect drug resistant organisms or treatment failures to first-line antimicrobials.

Urea breath test (UBT) has been approved by the Food and Drug Administration (FDA) for the detection of Helicobacter pylori. It is known that H. pylori possesses a urease enzyme that degrades urea in the stomach, producing carbon dioxide (CO (2)), which is then exhaled and can be detected in the lungs. Mycobacterium tuberculosis like H. pylori possesses a urease enzyme, which converts urea to carbon dioxide and ammonia. In a preclinical study, Jassal and colleagues demonstrated that TB-infected rabbits convert [(13)C]-labeled urea into [(13)C]-carbon dioxide ((13)CO(2)) in a matter of minutes. The (13)CO(2) in exhaled breath could be rapidly detected with an isotopic ratio mass spectrometer or a small ultraviolet (UV) absorbance spectrometer.

The primary objective of the current study is to evaluate the sensitivity and specificity of UBT in the diagnosis and treatment response of pulmonary TB. Secondary objectives are to assess the specificity of UBT for M. tuberculosis (UBT-TB) diagnosis in volunteers with and without H. pylori infection, examine the benefit of bismuth to make UBT-TB more specific for M. tuberculosis, and evaluate the correlation of the labeled (13)CO(2) signal with sputum colony forming unit (CFU) counts and the lower limit of signal detection versus CFU counts.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals (greater than or equal to18 years of age) are eligible to enter the study, if they meet the following criteria:

* Healthy volunteers (primary study group) or have a diagnosis of TB (as diagnosed by sputum smear tests; all three study groups).
* Willingness and ability to give informed consent.
* Willingness to undergo HIV testing.
* Willingness to have samples stored for future studies.

EXCLUSION CRITERIA:

Subjects are not eligible to enter the study, if they meet any of the following criteria:

* HIV infection.
* Past history of TB (Healthy volunteers only)
* Pregnancy and lactation
* Known history of diabetes
* Use of Tuberculosis treatment proton pump inhibitor treatments or use of bismuth containing preparations in the last 15 days prior to study entry.
* History of failed TB treatment
* Known allergy to aspirin or hypersensitivity to mannitol, citric acid or aspartame such as a clinical history suggestive of aminoacidurias.
* Any known medical disorder or other circumstance, which in the opinion of the PI, might make the participation of the individual unsafe or difficult. The reason for exclusion will be documented in the screening log.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2011-02-13; Study Completion 2016-03-30

CONTACTS AND LOCATIONS:
Overall Officials: Sophia B Siddiqui, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Unviersite de Bamako, Bamako, Mali

REFERENCES:
- [Background] Jassal M, Bishai WR. Extensively drug-resistant tuberculosis. Lancet Infect Dis. 2009 Jan;9(1):19-30. doi: 10.1016/S1473-3099(08)70260-3. Epub 2008 Nov 5. PMID 18990610
- [Background] Jassal MS, Nedeltchev GG, Lee JH, Choi SW, Atudorei V, Sharp ZD, Deretic V, Timmins GS, Bishai WR. 13[C]-urea breath test as a novel point-of-care biomarker for tuberculosis treatment and diagnosis. PLoS One. 2010 Aug 27;5(8):e12451. doi: 10.1371/journal.pone.0012451. PMID 20805989
- [Background] Bell GD, Weil J, Harrison G, Morden A, Jones PH, Gant PW, Trowell JE, Yoong AK, Daneshmend TK, Logan RF. 14C-urea breath analysis, a non-invasive test for Campylobacter pylori in the stomach. Lancet. 1987 Jun 13;1(8546):1367-8. doi: 10.1016/s0140-6736(87)90664-7. No abstract available. PMID 2884468